CLINICAL TRIAL: NCT02149654
Title: The Engager ALIGN Study. To Characterize the Safety and Clinical Benefit of the Engager Transcatheter Aortic Valve Implantation System in a Real World Environment.
Brief Title: Engager Align Post-market Clinical Study
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Organization: Medtronic Cardiovascular (Industry)
Other Study IDs: RAE00937
Record Dates: First submitted 2014-03-07; First posted 2014-05-29 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Aortic Valve Stenosis
Keywords: Transcatheter aortic valve implantation; Transcatheter aortic valve replacement; Engager transcatheter aortic valve implantation system; Engager bioprosthesis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Engager Transcatheter Aortic Valve Implantation System — The Engager Transcatheter Aortic Valve Implantation System is indicated for use in patients with symptomatic severe aortic valve stenosis requiring aortic valve replacement and are at high or extreme risk for operative mortality or comorbidity judged by the heart team to pose an absolute or relative contraindication for conventional aortic valve replacement. The system is intended for use in patients with a life expectancy of at least one year following TAVI. The intended performance of the system is to provide relief of aortic valve obstruction without inducing significant regurgitation, thereby restoring effective hemodynamic function of the diseased aortic valve. The intended purpose of the system in this clinical study is in line with the intended purpose in the Instructions for Use.

SUMMARY:
Purpose To characterize the safety and clinical benefit of the Engager Transcatheter Aortic Valve Implantation System in a real world environment.

Design Prospective non-randomized, non-interventional, multicenter, single-arm, post-market study.

250 Patients will have the Engager bioprosthesis implanted. Patients will be followed at 1 month, 6 months, and 12 months after the procedure. The recruitment period will be approximately 12 months, so the total study duration will be 24 months.

DETAILED DESCRIPTION:
The study objective is to characterize the safety and clinical benefit of the Engager Transcatheter Aortic Valve Implantation System in a real world setting.

The primary endpoint of this study is all-cause mortality at 30 days or during index hospitalization.

Secondary endpoints of this study are:

* Device success according to VARC2 is defined as:
* absence of procedural mortality (all-cause mortality at discharge, 30 days or during index hospitalization), AND
* correct positioning of the Engager bioprosthesis in the proper anatomic location, AND
* Engager bioprosthesis performing as intended (no prosthesis-patient mismatch and mean aortic valve gradient < 20 mmHg or peak velocity < 3 m/s, AND no moderate or severe regurgitation).
* Composite early safety (at 30 days) according to VARC2 includes the following components:
* all-cause mortality
* all stroke
* life-threatening bleeding
* acute kidney injury (stage 2-3)
* coronary artery obstruction requiring intervention
* major vascular complication
* valve-related dysfunction requiring repeat procedure (BAV, TAVI or SAVR)
* Clinical efficacy according to VARC2 at 6 months and 1 year is defined as:
* all-cause mortality
* all stroke
* hospitalizations for valve-related symptoms or worsening congestive heart failure (CHF)
* NYHA class III or IV
* valve-related dysfunction (mean aortic valve gradient ≥20 mm Hg, effective orifice area (EOA) ≤0.9-1.1 cm² and/or Doppler velocity index (DVI) <0.35 m/s, AND/OR moderate or severe prosthetic valve regurgitation)
* Time-related valve safety accordingly to VARC2 at 6 months and 1 year is defined as:
* Structural valve deterioration
* Valve-related dysfunction (mean aortic valve gradient ≥20 mm Hg, (EOA) ≤0.9-1.1 cm² and/or (DVI) <0.35 m/s, AND/OR moderate or severe prosthetic valve regurgitation)
* Requiring repeat procedure (TAVI or SAVR)
* Prosthetic valve endocarditis
* Prosthetic valve thrombosis
* Thrombo-embolic events (e.g. stroke)
* VARC bleeding, unless clearly unrelated to valve therapy (e.g. trauma)

  * All-cause mortality at 6 months and 1 year
  * Cardiovascular mortality at 30 days, 6 months and 1 year
  * Incidence of TAVI-related complications at 30 days, 6 months and 1 year:
* Myocardial infarction
* Periprocedural and spontaneous stroke
* Life-threatening, major and minor bleedings
* Acute kidney injury state 1, 2 and 3
* Apical and vascular complications
* Conduction disturbances
* Conversion to open-heart surgery
* Unplanned use of cardiopulmonary bypass
* Coronary obstruction and dissection
* Ventricular septal perforation
* Mitral valve apparatus damage or dysfunction
* Cardiac tamponade
* Endocarditis
* Valve thrombus
* Valve migration, embolization or ectopic valve deployment
* Valve in valve deployment

  * Total, transvalvular and paravalvular regurgitation as measured by TTE at 30 days and 1 year
  * Mean aortic valve gradient, peak velocity and effective orifice area as measured by TTE at 30 days and 1 year
  * Engager implant depth as measured by standard of care angiography at the end of implant procedure
  * Incidence and rationale for permanent pacemaker implantation after Engager implant procedure
  * Changes in Quality of Life as measured by the EQ5D questionnaire at baseline, discharge, 30 days, 6 months and 1 year
  * Length of stay during index hospitalization (ICU and general ward)
  * Incidence of re-hospitalization at 30 days, 6 months and 1 year

Subject population All patients with severe aortic stenosis requiring treatment, who are selected by a heart team to be treated electively with the Engager Transcatheter Aortic Valve Implantation System are eligible to be included in this study.

Treatment The Engager Transcatheter Aortic Bioprosthesis will be implanted using the Engager Transcatheter Delivery System. The bioprosthesis is delivered transapically on a catheter during a beating heart procedure.

ELIGIBILITY:
Inclusion Criteria:

Patient can be included if ALL of the following criteria are met:

* Patient with severe aortic valve stenosis requiring treatment;
* Patient is an acceptable candidate for elective treatment with the Medtronic Engager Transcatheter Aortic Valve Implantation System and in conformity with the local regulatory requirements;
* Patient is above the minimum age as required by local regulations to be participating in a clinical study;
* The patient has been informed of the nature of the study and has consented to participate, and has authorized the collection and release of his/her medical information by signing a consent form (Patient Informed Consent Form or Data Release Form).

Exclusion Criteria:

Patient will not be included if any of the following conditions exist:

* Known hypersensitivity or contraindication to aspirin, heparin, ticlopidine, clopidogrel, Nitinol of contrast medium that cannot be adequately controlled with pre-medication;
* Intracardiac mass, thrombus, or vegetation;
* Aortic aneurysm;
* Sepsis or acute endocarditis;
* Bleeding diathesis, or coagulopathy;
* Cardiogenic shock, suspected cardiogenic shock;
* Unicuspid or bicuspid aortic valve;
* Pre-existing prosthetic heart valve in aortic position;
* Patient is currently enrolled in another investigational device or drug trial;
* Patients with life expectancy less than 12 months after TAVI.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with severe aortic stenosis requiring treatment, who are selected by a heart team to be treated electively with the Engager Transcatheter Aortic Valve Implantation System are eligible to be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
is to characterize the safety and clinical benefit of the Engager Transcatheter Aortic Valve Implantation System in a real world setting. | 12 months
  The study objective is to characterize the safety and clinical benefit of the Engager Transcatheter Aortic Valve Implantation System in a real world setting.
  The primary endpoint of this study is all-cause mortality at 30 days or during index hospitalization.

SECONDARY OUTCOMES:
Device success according to VARC2 | 12 Month follow up
  Absence of procedural mortality (all-cause mortality at discharge, 30 days or during index hospitalization), AND correct positioning of the Engager bioprosthesis in the proper anatomic location, AND Engager bioprosthesis performing as intended (no prosthesis-patient mismatch and mean aortic valve gradient < 20 mmHg or peak velocity < 3 m/s, AND no moderate or severe regurgitation).
  Composite early safety (at 30 days) according to VARC2. All-cause mortality at 6 months and 1 year; Cardiovascular mortality at 30 days, 6 months and 1 year; Incidence of TAVI-related complications at 30 days, 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik Treede, MD, Principal Investigator — Universitätsklinikum Hamburg
Locations (1):
- Medtronic Bakken Research Center, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided